CLINICAL TRIAL: NCT01567969
Title: Family Health and Development Project: Intensive In-home Child and Adolescent Psychiatric Service (IICAPS) vs. Home-based Child Treatment Coordination (Home-based CTC) for Seriously Emotionally Disturbed Children
Brief Title: Family Health and Development Project
Acronym: FHDP
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1102008073
Record Dates: First submitted 2012-03-12; First posted 2012-03-30 (Estimated); Last update posted 2016-10-14 (Estimated); Status verified 2016-10

CONDITIONS: Serious Emotional Disturbance
Keywords: mental health services; child behavior disorders; child psychiatry
MeSH Terms: conditions — Child Behavior Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- IICAPS (Experimental): Provision of Intensive In-home Child and Adolescent Psychiatric Service, a six to seven month family-focused in-home psychiatric intervention.
  Interventions: Behavioral: Intensive In-home Child and Adolescent Psychiatric Service
- Home-based CTC (Active Comparator): Provision of Home-based Child Treatment Coordination, a six to seven month child-focused case management service with monthly in-home visits with the child's parent/legal guardian.
  Interventions: Behavioral: Home-based Child Treatment Coordination

INTERVENTIONS:
Behavioral: Intensive In-home Child and Adolescent Psychiatric Service — A six to seven month intensive intervention provided by a clinical team consisting of a master's-level clinician and a bachelor's-level mental health counselor delivering comprehensive psychiatric and case management services in the child's home. One or both members of the team works with the child and the family three times a week in the home. Delivery of direct and indirect services average 5.5 hours of service per week.
  Arms: IICAPS
Behavioral: Home-based Child Treatment Coordination — A six to seven month home-based case management service delivered by a master's level clinician. The coordinator meets with the child's parent/legal guardian in the child's home once a month and conducts weekly phone conversations to facilitate referral and access to appropriate mental health services for the child.
  Arms: Home-based CTC

SUMMARY:
The Family Health and Development Project (FHDP) is a randomized controlled trial to evaluate the effectiveness of the Intensive In-home Child and Adolescent Psychiatric Service (IICAPS) intervention, targeting emotionally, behaviorally, and/or psychiatrically disordered children at risk of a psychiatric inpatient admission and their families. Children and families are randomized to receive IICAPS or Home-based Child Treatment Coordination (Home-based CTC), a home-based case management intervention for coordination of mental health services for children. Approximately 144 children and their families will be enrolled for a 12 month study period. Data will be collected through interviews with the child's parent/legal guardian, and from the child's teacher, the child's school, and the Department of Social Services (claims data). This study will test the hypotheses that children receiving IICAPS will be less likely to exhibit out-of-control behaviors and less likely to experience a psychiatric hospitalization and/or out-of-home placement during and up to six months post-discharge from services.

DETAILED DESCRIPTION:
The Family Health and Development Project (FHDP) is a randomized controlled trial to evaluate the effectiveness of the Intensive In-home Child and Adolescent Psychiatric Service (IICAPS) intervention, targeting emotionally, behaviorally, and/or psychiatrically disordered children at risk of a psychiatric inpatient admission and their families. Children and families are randomized to receive IICAPS or Home-based Child Treatment Coordination (Home-based CTC), a home-based case management intervention for coordination of mental health services for children. Approximately 144 children and their families will be enrolled for a 12 month study period. Each study intervention is six to seven months in duration, with approximately 6 additional months of follow-up.

Data are collected from the identified child's parent/legal guardian during three in-person assessment interviews (at enrollment, at end of study treatment, and at 12-months), and during brief monthly phone interviews. Data are collected on child psychiatric symptoms and behavior, child psychiatric inpatient admissions and other service utilization, parenting practices, and parental problem solving skills. Additional data are collected from the child's teacher (child's behavior at school) and the child's school (days missed, suspensions, expulsions, disciplinary action) at baseline, 6-months, and 12-months. Service utilization data will be collected from the Connecticut Department of Social Services using claims data.

The main study aim is to evaluate the efficacy of IICAPS for youth with serious and pervasive mental health problems that places them at risk for institutional placement, and test the hypotheses that children receiving IICAPS will be less likely to exhibit out-of-control behaviors and less likely to experience a psychiatric hospitalization and/or out-of-home placement during and up to six months post-discharge from services. The second study aim is to evaluate how the efficacy of IICAPS for youth with serious and pervasive mental health problems is achieved, with specific focus on parenting practices, parental problem solving techniques, and parental perception of the child.

ELIGIBILITY:
Inclusion Criteria:

* child has a Diagnostic and Statistical Manual-IV (DSM-IV) diagnosis
* child at risk of psychiatric hospitalization due to serious out-of-control behaviors
* child resides in home of legal guardian, who is primary caregiver
* child insured by Medicaid
* score in the borderline clinical or clinical range on the Externalizing Scale of the Child Behavior Checklist (CBCL)

Exclusion Criteria:

* referred to IICAPS by a probation officer
* suffers from an unstable, chronic medical comorbidity
* prior receipt of IICAPS

Ages: 6 Years to 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 110 (Actual)
Dates: Start 2011-05; Primary Completion 2015-11 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in Child Out-of-control Behavior | Baseline up to 7 months post-baseline
  Child out-of-control behavior is measured by the Retrospective Modified Overt Aggression Scale (R-MOAS). This instrument is administered at baseline and at the end of study treatment (IICAPS or Home-based CTC), at approximately 6 to 7 months post-baseline.
Change in Child Out-of-control Behavior | Baseline to 12 months post-baseline
  Child out-of-control behavior is measured by the Retrospective Modified Overt Aggression Scale (R-MOAS). This instrument is administered at baseline and at the 12 months post-baseline.
Change in Child Out-of-control Behavior | Up to 12 months post-baseline
  Child out-of-control behavior is measured by the Retrospective Modified Overt Aggression Scale (R-MOAS) monthly from baseline to 12-months post-baseline.
Change in Child Psychiatric Inpatient Admissions and Days | Baseline (measure of prior 6 months) up to 7 months post-baseline (measuring time since baseline)
  Child psychiatric inpatient admissions and days will be collected for the six-months prior to study enrollment, and measured against child psychiatric inpatient admissions and days from baseline to the end of the study treatment intervention (IICAPS or Home-based CTC), at approximately 6 to 7 months post-baseline.
Change in Child Psychiatric Inpatient Days and Admissions | Baseline (measure of 6 months prior) to 12 months post-baseline
  Child psychiatric inpatient admissions and days will be collected for the six-months prior to study enrollment, and measured against child psychiatric inpatient admissions and days from baseline to 12 months post-baseline.
Change in Child Out-of-control Behavior | Baseline up to 7 months post-baseline
  Child out-of-control behavior as measured by the Child Behavior Checklist (CBCL). This instrument is administered at baseline and at the end of study treatment (IICAPS or Home-based CTC), at approximately 6 to 7 months post-baseline.
Change in Child Out-of-control Behavior | Baseline to 12 months post-baseline
  Child out-of-control behavior as measured by the Child Behavior Checklist (CBCL). This instrument is administered at baseline and at 12 months post-baseline.

SECONDARY OUTCOMES:
Change in Parenting Practices | Baseline up to 7 months post-baseline
  Parenting practices will be measured using the Alabama Parenting Questionnaire (APQ)administered at baseline and at the end of the study treatment intervention (IICAPS or Home-based CTC).
Change in Parenting Practices | Baseline to 12 months post-baseline
  Parenting practices will be measured using the Alabama Parenting Questionnaire (APQ)administered at baseline and at 12-months post-baseline.
Change in Parental Problem Solving | Baseline up to 7 months post-baseline
  Parental problem solving will be measured using the Problem Solving subscale of McMaster Family Assessment Device (FAD) administered at baseline and at the end of the study treatment intervention (IICAPS or Home-based CTC).
Change in Parental Problem Solving | Baseline to 12 months post-baseline
  Parental problem solving will be measured using the Problem Solving subscale of McMaster Family Assessment Device (FAD) administered at baseline and at 12-months post-baseline.
Change in Parental Perception of their Child | Baseline up to 7 months post-baseline
  Parental perception of their child will be measured using the Parent Cognition Scale (PCS) administered at baseline and at the end of the study treatment intervention (IICAPS or Home-based CTC).
Change in Parental Perception of their Child | Baseline to 12 months post-baseline
  Parental perception of their child will be measured using the Parent Cognition Scale (PCS) administered at baseline and at 12-months post-baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Joseph L. Woolston, M.D., Principal Investigator — Yale University
Locations (1):
- Yale University Child Study Center, New Haven, Connecticut, United States

REFERENCES:
- [Background] Woolston JL, Adnopoz JA, Berkowitz SJ. IICAPS: A Home-Based Psychiatric Treatment for Children and Adolescents. New Haven: Yale University Press, 2007.